CLINICAL TRIAL: NCT02603497
Title: Pharmacokinetic (PK) Study of ASP015K -Evaluation of Pharmacokinetics in Patients With Impaired Renal Function and Subjects With Normal Renal Function-
Brief Title: Pharmacokinetics Study in Patients With Impaired Renal Function and Subjects With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 015K-CL-PK11
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2019-04

CONDITIONS: Patients With Impaired Renal Function
Keywords: ASP015K; impaired renal function; Pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency | interventions — peficitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Subjects with normal renal function) (Experimental): Oral
  Interventions: Drug: ASP015K
- Mild renal impairment (Experimental): Oral
  Interventions: Drug: ASP015K
- Moderate renal impairment (Experimental): Oral
  Interventions: Drug: ASP015K
- Severe renal impairment (Experimental): Oral
  Interventions: Drug: ASP015K

INTERVENTIONS:
Drug: ASP015K — oral

SUMMARY:
The objective of this study is to compare the pharmacokinetics of ASP015K in patients with impaired renal function and subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

All subject

* Body weight): ≥40.0 kg and <90.0 kg
* Body mass index BMI: ≥17.6 and <30.0
* Female subject must either:

  * Be post-menopausal or surgically sterile.
  * Agree not to try to become pregnant starting at the time of informed consent throughout the study period and for 60 days after the final study drug administration if she is of childbearing potential.
* Female subjects who agree not to breastfeed starting at informed consent and throughout the study period and for 60 days after the final study drug administration
* Agree not to donate ova for female / sperm for male starting at informed consent and throughout the study period and for 60/90 days after the final study drug administration
* Agree to use highly effective contraception

Patients with impaired renal function

* Patients with eGFR by GFR predictive equation for Japanese within the following ranges at screening and who is not undergoing dialysis.

  * Patients with mild impaired renal function (eGFR; ≥60 mL/min/1.73 m2 and <90 mL/min/1.73 m2)
  * Patients with moderate impaired renal function (eGFR; ≥30 mL/min/1.73 m2 and <60 mL/min/1.73 m2)
  * Patients with severe impaired renal function (eGFR; ≥15 mL/min/1.73 m2 and <30 mL/min/1.73 m2)
* Patients whose treatment regimen (including diet) for renal impairment or complications remain unchanged within 14 days prior to hospital admission day (Day -1), or patients who receive treatments (including diet) that need not to be changed during the period from 14 days before hospital admission day (Day -1) to follow-up examination in the opinion of the investigator or sub-investigator.

Subjects with normal renal function

* Subjects with eGFR by GFR predictive equation for Japanese ≥ 90 mL/min/1.73 m2 at screening
* Subjects who is healthy, as judged by the investigator or sub-investigator based on physical examinations (subjective symptoms and objective findings) and all tests obtained at screening and during the period from hospital admission to immediately before study drug administration

Exclusion Criteria:

All subjects

* Received or is scheduled to receive any study drugs in other clinical trials or post-marketing studies within 120 days before screening or during the period from screening to the hospital admission day (Day -1)
* Deviate from the following provided range of blood pressure, pulse rate, body temperature and standard 12-lead ECG at screening or the hospital admission day (Day -1)
* Subjects who meet any of the criteria for laboratory tests at screening or the hospital admission day (Day -1). Normal ranges of each test specified at the study site or the test/assay organization will be used as the normal ranges in this study.
* Complication or history of drug allergies
* Developed upper gastrointestinal symptoms within 7 days before the hospital admission day (Day -1)
* Complication or history of hepatic disease
* Complication of long QT syndrome, congenital short QT syndrome
* A history of gastrointestinal resection
* Subjects with a complication or history of endocrine disease
* Subjects with a complication or history of malignant tumor
* Subjects with a complication or history of lymphatic disease
* Applies to any of following concerns of tuberculosis

  * A history of active tuberculosis
  * Abnormalities detected on a chest X-ray test (at screening)
  * Contact with infectious tuberculous patients
* Applies to any of following concerns, with regard to infection except for tuberculosis

  * A complication or history of severe herpes zoster or herpes zoster disseminated
  * At least twice of relapse of localized herpes zoster
  * Inpatient hospital care for severe infectious diseases within 90 days before the hospital admission day (Day -1)
  * Treatment with intravenous antibiotics within 90 days before the hospital admission day (Day -1) (prophylactic antibiotics are not applicable).
  * Other than above, a subject with a high risk of developing infectious disease (e.g. subjects with urethral catheterisation) in judgment of the investigator or sub-investigator.
* Vaccination of live vaccines or live attenuated vaccines within 56 days before the hospital admission day (Day -1) (Inactivated vaccines such as influenza vaccine and pneumococcal vaccine are not applicable.)
* A history of clinically serious allergies
* Previously received administration of ASP015K
* Excessive alcohol drinking or smoking

Patients with impaired renal function

* Patients who received or are scheduled to receive any new drugs within 14 days before the hospital admission day (Day -1)
* Patients who receive dialysis, or received renal transplantation
* Patients who developed acute changes in renal function and in all laboratory test results within 28 days before screening and patients with impaired renal function who may need new concomitant therapies during the study period.
* Patients with a complication of severe heart disease, NYHA class III or IV cardiac failure.
* Complication of alimentary disease, cerebrovascular disorder, respiratory disease
* Patients with tubular dysfunction, obvious urination impaired

Subjects with normal renal function

* Subjects who received or is scheduled to receive medications (including over-the-counter [OTC] drugs) within seven days before the hospital admission day (Day -1).
* Subjects with a complication or history of heart disease, respiratory disease, alimentary disease, renal disease, endocrine disease, urological disease, cerebrovascular disorder

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) parameter of ASP015K: AUCinf | pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
  AUCinf: Area under the concentration-time curve from the time of dosing extrapolated to time infinity
PK parameter of ASP015K: Cmax | pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
  Cmax: Maximum concentration
PK parameter of metabolites: AUCinf | pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
PK parameter of metabolites: Cmax | pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
Safety assessed by Adverse Events (AEs) | Up to 7 days after the study drug dosing
Safety assessed by Vital signs | Up to 7 days after the study drug dosing
  Supine blood pressure, supine pulse rate and axillary body temperature
Safety assessed by Laboratory tests | Up to 7 days after the study drug dosing
  Hematology, blood biochemistry and urinalysis
Safety assessed by 12-lead ECGs | Up to 7 days after the study drug dosing
  ECG: Electrocardiogram

SECONDARY OUTCOMES:
PK parameters of ASP015K: AUClast | pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
  AUClast: Area under the concentration-time curve from the time of dosing extrapolated to the last measurable concentration
PK parameters of ASP015K: t1/2 | pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
  t1/2: Terminal elimination half-life
PK parameters of ASP015K: tmax | pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
  tmax: Time of Cmax
PK parameters of ASP015K: CL/F | pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
  CL/F: Apparent total systemic clearance
PK parameters of ASP015K: Vz/F | pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
  Vz/F: Apparent volume of distribution during the terminal elimination phase
PK parameters of metabolites: AUClast | pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
PK parameters of metabolites: t1/2 | pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
PK parameters of metabolites: tmax | pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (2):
- Japan (2):
  - Site JP00001, Tokyo
  - Site JP00002, Tokyo

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Toyoshima J, Shibata M, Kaibara A, Kaneko Y, Izutsu H, Nishimura T. Population pharmacokinetic analysis of peficitinib in patients with rheumatoid arthritis. Br J Clin Pharmacol. 2021 Apr;87(4):2014-2022. doi: 10.1111/bcp.14605. Epub 2020 Dec 1. PMID 33068028
- [Derived] Miyatake D, Shibata T, Shibata M, Kaneko Y, Oda K, Nishimura T, Katashima M, Sekino H, Furihata K, Urae A. Pharmacokinetics and Safety of a Single Oral Dose of Peficitinib (ASP015K) in Japanese Subjects with Normal and Impaired Renal Function. Clin Drug Investig. 2020 Feb;40(2):149-159. doi: 10.1007/s40261-019-00873-7. PMID 31729626